CLINICAL TRIAL: NCT02384824
Title: Evaluation of Delayed Plaque Morphology by Optical Coherence Tomography (OCT) in Patients With Acute ST Segment Elevated Myocardial Infarction (STEMI) After Thrombus Aspiration During Primary Percutaneous Intervention (PCI)
Brief Title: Delayed Plaque Morphology in Patients With STEMI After Thrombus Aspiration During Primary PCI
Acronym: STEMI-OCT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jian'an Wang,MD,PhD (Other)
Responsible Party: Sponsor-Investigator, Jian'an Wang,MD,PhD, President of Second Affiliated Hospital, School of Medicine, Zhejiang University & Chief of Cardiology, Second Affiliated Hospital, School of Medicine, Zhejiang University
Organization: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Other Study IDs: SAHZJU CT003
Record Dates: First submitted 2015-01-15; First posted 2015-03-10 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Coronary Artery Disease; Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Primary Percutaneous Intervention — angiography, manual aspiration thrombectomy and antiplatelet therapy

SUMMARY:
The purpose of this study is to characterize the plaque morphology in patients with acute STEMI by OCT after aspiration thrombectomy.

DETAILED DESCRIPTION:
Current guideline for treating acute STEMI is primarily PCI and stent placement in the infarct-related coronary artery. But, the underlying plaque morphology is not routinely identified due to the limited resolution of conventional imagine modalities. However, autopsy studies have shown that there are different atherosclerotic plaque morphologies involving in acute thrombotic occlusion of coronary arteries other than atherosclerotic plaque rupture, such as plaque erosion, calcified nodule, etc. Some studies have suggested that PCI and stenting might not always be necessary in about 30 - 40% of ACS patients, and an alternative treatment strategy is needed for these patients based on the characteristics of plaque morphology.

100 subjects who meet the inclusion/exclusion criteria will undergo emergent angiography and followings: If no thrombus was observed, OCT examination will be performed in the target vessel;

If thrombosis was confirmed, the subject will undergo manual aspiration thrombectomy and antiplatelet therapy, and TIMI flow will be assessed:

If TIMI flow grade < 3, the subject will receive stent implantation as the standard of care followed by OCT examination; If TIMI flow grade of 3, the subject will not receive stent implantation but will be sent to CCU for monitoring and antiplatelet treatment, and have a repeat angiography and OCT examination at Day 7; within the 7days post STEMI, ischemia-driven angiography and/or PCI are allowed, and an OCT examination will be performed in these subject before PCI.

Patients without undergoing initial stent implantation will have scheduled 30-day and 12-month follow-ups for clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical inclusion criteria:

   * Age > 18 years
   * Onset of STEMI > 30 minutes, but < 12 hours
   * ST segment elevation in at least 2 contiguous leads of≥ 1mm or newly developed LBBB on ECG
   * Willing and able to provide informed consent
2. Angiographic inclusion criteria:

   * Having at least one infarct-related coronary artery, of which
   * The Culprit lesion is suitable for stenting;
   * The reference diameter of culprit vessel is ≥ 2.5 mm but ≤ 4 mm;
   * The TIMI flow is ≤ 1 in culprit lesion segment prior to guide wire crossing
   * No excessive tortuosity and calcification in the culprit lesion segment that allowing stent implantation

Exclusion Criteria:

1. Clinical exclusion criteria:

1. Contraindicating to any concomitant study medications
2. Having cardiogenic shock with hemodynamic instability
3. A history of bleeding diathesis or known coagulopathy
4. A history of cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months; or a history of intracranial tumor, aneurysm or arteriovenous malformations; or a history of active peptic ulcer or active gastrointestinal (GI) bleeding within the past 2 months; or planned major procedure within 6 weeks; or known platelet count < 100,000 /mm3 or Hb < 10 g/dL
5. Planned surgery which may cause discontinuation of ADP-receptor antagonist
6. Other serious illness (e.g., cancer) that may reduce life expectancy to less than 1 year
7. Repeated MI within 7 days of hospitalization for acute MI

   * Angiographic exclusion criteria:

     * Bifurcated lesion unable to identify the culprit lesion
     * The culprit lesion is located in the left main artery
     * Diffusive lesions without distinguishable culprit lesion
     * Previous stent implantation in the culprit lesion segment or STEMI caused by stent thrombosis
     * Likely CABG procedure within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acute STEMI
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
plaque morphology by OCT | at the 7th day post PCI/aspiration thrombectomy

SECONDARY OUTCOMES:
Re-hospitalization due to cardiac symptoms | 30 days & 12 months
Myocardial infarction related to the target vessel | 30 days & 12 months